CLINICAL TRIAL: NCT01849588
Title: A Prospective Study of HCV-RNA Kinetics During Treatment With Sorafenib in Patients With Advanced Hepatocellular Carcinoma and Chronic Hepatitis C
Brief Title: HCV-RNA Kinetics During Sorafenib for Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-213
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Hepatocellular Cancer
Keywords: Hepatitis C positive
MeSH Terms: conditions — Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Sorafenib taken orally twice per day
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib
  Other Names: Nexavar

SUMMARY:
This research study is a Phase IV clinical trial. Phase IV trials are used to further test and monitor the safety of a drug approved by the FDA and to see if the drug has any other indications that can be used to treat different diseases.

Sorafenib is a new drug, which is approved under the brand name Nexavar for the treatment of liver cancer. It is also currently being tested in various other cancers. Sorafenib works by slowing down and/or stopping the development of new cancer cells and new blood vessels. By slowing down and/or stopping the growth of new blood vessels around a tumor, it is believed that sorafenib prevents or slows down the growth of tumors.

The researchers of this study would like to study the effects of sorafenib on hepatitis C by drawing additional research blood samples from people infected with hepatitis C who are receiving sorafenib treatment for liver cancer. These tests will measure certain proteins in the blood (HCV-RNA) which may indicate if sorafenib has any effect on the hepatitis C virus.

DETAILED DESCRIPTION:
This is a prospective, open-label, non-interventional trial to evaluate HCV-RNA levels during treatment with Sorafenib in patients with advanced hepatocellular carcinoma.

Participants will receive Sorafenib 400mg orally twice daily. HCV-RNA (Hepatitis C Virus - Ribonucleic Acid) levels will be measured at baseline, week 2 of sorafenib, week 4 of sorafenib, week 6 of sorafenib, week 8 of sorafenib, week 12 of sorafenib, and 2 weeks after discontinuing sorafenib. HCV-RNA levels will be measured by drawing about 2 tablespoons of blood

During the study period, tumor assessments will be done by MRI (magnetic resonance imaging) or CT (computed tomography) scans at baseline and every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or radiologically confirmed advanced HCC
* Detectable HCV RNA with anti-HCV-positivity
* Life expectancy of at least 3 months
* Willing to use adequate contraception

Exclusion Criteria:

* Pregnant or breastfeeding
* Undetectable HCV RNA
* Uncontrolled hypertension
* Active or clinically significant cardiac disease
* Thrombolic, embolic, venous or arterial events within 6 months of informed consent
* Pulmonary hemorrhage/bleeding event (NCI-CTCAE grade 2 or higher) within 4 weeks before study entry
* Previously untreated or concurrent cancer except cervical cancer in situ, treated basal cell carcinoma or superficial bladder tumor
* Presence of non-healing wound, ulcer or bone fracture
* History of organ allograft
* Known or suspected allergy or hypersensitivity to any of the study drugs
* Any malabsorption condition
* Inability to comply with the protocol and/or not willing or not available for follow up
* Major surgery within 30 days prior to start of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zhu, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between December 2013 and December 2015
Groups:
- Sorafenib: Sorafenib taken orally twice per day
  Sorafenib
Period: Overall Study
Arm/Group | Sorafenib
Started | 3
Completed | 0
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 57.8 [56.9 to 61.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Decline in HCV-RNA Level
Description: Successful decline in HCV (hepatitis C virus)-RNA level, with success defined as a decrease of at least two logs of HCV-RNA between baseline and any subsequent measurement.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm: Sorafenib taken orally twice per day
  Sorafenib
Arm/Group | Treatment Arm
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Time to Radiological Tumor Progression
Description: Time to radiological tumor progression is defined as the time period between enrollment and the earlier of tumor progression and death. Participants who are alive and progression-free at the date of last contact will be censored at this date.
Time Frame: 2 years
Population: Study was terminated early due to slow accrual.
Measure: Mean (Full Range); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 3
months | 5.68 [1.84 to 12.43]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time period between enrollment and the date of death. Participants who are still alive at last contact will be censored at this date.
Time Frame: 2 years
Measure: Mean (Full Range); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 3
months | 8.36 [2.76 to 13.65]

4. Other Pre Specified Outcome: Decrease Alpha-fetoprotein(AFP) Level > 20% From the Baseline
Description: The proportion of participants with a decrease of greater than 20% in AFP (alpha-fetoprotein) level between baseline and any subsequent measurement following treatment with sorafenib will be reported.
Time Frame: 2 years
Population: AFP levels were not available for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Participants are monitored for adverse events throughout their entire time on study. This was a maximum of 13 months.
Description: Only events possibly, probably, or definitely related to administration of sorafenib are listed here.
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=3)
diarrhea (Gastrointestinal disorders) | 3
fatigue (General disorders) | 2
palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 2
nausea (Gastrointestinal disorders) | 2
platelet count decreased (Investigations) | 3
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
anorexia (Metabolism and nutrition disorders) | 1
erythema (Skin and subcutaneous tissue disorders) | 1
GI bleed (Gastrointestinal disorders) | 1
low phosphorus (Metabolism and nutrition disorders) | 3
elevated bilirubin (Investigations) | 3
elevated alkaline phosphatase (Investigations) | 3
hypertension (Vascular disorders) | 1
facial rash (Skin and subcutaneous tissue disorders) | 1
vomiting (Gastrointestinal disorders) | 1
weight loss (Investigations) | 1
abdominal pain (Gastrointestinal disorders) | 1
bloating (Gastrointestinal disorders) | 2
anemia (Blood and lymphatic system disorders) | 2
anxiety (Psychiatric disorders) | 1
ascites (Gastrointestinal disorders) | 1
chills (General disorders) | 1
dyspepsia (Gastrointestinal disorders) | 1
periodontal disease (Gastrointestinal disorders) | 1 — gum bleeding
headache (Nervous system disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 2
hyperkalemia (Metabolism and nutrition disorders) | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 1
hypocalcemia (Metabolism and nutrition disorders) | 1
hypoglycemia (Metabolism and nutrition disorders) | 1
hypomagnesemia (Metabolism and nutrition disorders) | 1
hyponatremia (Metabolism and nutrition disorders) | 1
non-cardiac chest pain (General disorders) | 1
pruritis (Skin and subcutaneous tissue disorders) | 1
SGOT increased (Investigations) | 3
SGPT increased (Investigations) | 2

LIMITATIONS AND CAVEATS:
Study was terminated early due to slow accrual, therefore a small number of participants were analyzed and the data are not statistically significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No